CLINICAL TRIAL: NCT04043988
Title: Management of Diverticulitis in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, David A. Talan, Principal Investigator, Olive View-UCLA Education & Research Institute
Other Study IDs: 1396802
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to describe current treatment practices in the US for managing acute uncomplicated diverticulitis. In addition, we will identify clinical factors associated with the decision to discharge versus hospitalize patients with uncomplicated diverticulitis with the goal of informing clinical decision-making and providing a foundation for diagnostic algorithms to guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Emergency department presumptive or confirmed final diagnosis of acute diverticulitis
* Verbal or written consent provided in English (or Spanish depending on study site)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency departments at EMERGEncy ID NET sites will be screened for study eligibility by study coordinators or treating clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 718 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Rates of hospital admission | Day 1
  Rates of hospital admission from the emergency department among patients being treated for acute diverticulitis will be determined. In addition, factors associated with hospital admission will be examined.
Rate of Imaging | Day 1
  The rate of imaging performed in the emergency department among patients treated for acute diverticulitis will be determined. Factors associated with imaging will also be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Olive View-UCLA Medical Center, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: No